CLINICAL TRIAL: NCT07296172
Title: Surgical Difficulty and Operation Time as Determinants of Outcomes in Mandibular Third Molar Surgery
Brief Title: Difficulty, Time & M3 Surgery Outcomes
Status: Completed | Type: Observational
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Dilara KAZAN, assistant prof, Bahçeşehir University
Other Study IDs: GO 15/556
Record Dates: First submitted 2025-11-26; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Third Molar Extraction Surgery; Third Molar Impaction; Satisfaction Survey

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing surgical extraction of impacted mandibular third molars

SUMMARY:
This prospective observational cohort study is designed to evaluate early postoperative complications and patient-reported satisfaction following surgical extraction of impacted mandibular third molars under local anesthesia in adult patients. Standardized surgical and postoperative protocols are applied to all participants. The primary objective is to assess overall patient satisfaction on postoperative day 7 using a structured questionnaire. Secondary objectives are to describe the frequency and characteristics of early postoperative pain, swelling, trismus and other complications in the first postoperative week after surgery.

DETAILED DESCRIPTION:
Adult patients requiring surgical removal of an impacted mandibular third molar under local anesthesia will be prospectively enrolled at a single oral and maxillofacial surgery center. All procedures will be performed using a standardized surgical technique and a uniform postoperative medication and care protocol. Clinical examinations and patient-reported outcome measures will be obtained at baseline and at the postoperative day-7 follow-up visit. The study focuses on describing the early postoperative course after third molar surgery and on exploring how early complications relate to overall patient satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of one impacted mandibular third molar indicated for surgical extraction
* Surgical removal of the impacted mandibular third molar planned under local anesthesia
* Good general health (ASA I-II)
* Ability to understand the study information and provide written informed consent
* Willingness and ability to attend the postoperative day-7 follow-up visit and to complete all study questionnaires

Exclusion Criteria:

* Systemic diseases corresponding to ASA III or higher
* Acute infection at the surgical site (e.g. acute pericoronitis, abscess) requiring emergency treatment
* Previous surgical intervention at the same mandibular third molar region
* Pregnancy or lactation
* History of radiotherapy or chemotherapy involving the head and neck region
* Known bleeding disorders or current use of anticoagulant medication that cannot be safely modified for surgery
* Chronic use of systemic corticosteroids, immunosuppressive drugs, or long-term analgesic therapy that may interfere with pain assessment or healing
* Known allergy or contraindication to the local anesthetic or routinely used postoperative medications in this study
* Significant cognitive or psychiatric disorders, or language barriers that prevent reliable completion of the questionnaires

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients referred to the Department of Oral and Maxillofacial Surgery at Hacettepe University for surgical removal of an impacted mandibular third molar under local anesthesia. Eligible participants are generally healthy (ASA I-II), present with a single impacted mandibular third molar indicated for extraction, and are able to attend the postoperative day-7 follow-up visit and complete all study questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Total score on a 20-item postoperative patient satisfaction questionnaire following surgical extraction of impacted mandibular third molars | day 7
  Patient satisfaction will be assessed on postoperative day 7 using a 20-item postoperative mandibular third molar surgery patient satisfaction questionnaire. The questionnaire evaluates domains such as pain control, swelling, mouth opening, intraoperative and postoperative comfort, information provided by the surgeon, ability to chew and perform daily activities, willingness to undergo the procedure again, and overall satisfaction with care. Each item is rated on a 5-point Likert-type scale (1 = lowest satisfaction, 5 = highest satisfaction). A total satisfaction score will be calculated by summing all item scores, resulting in a minimum total score of 20 and a maximum total score of 100.

SECONDARY OUTCOMES:
Incidence and severity of early postoperative complications after surgical extraction of impacted mandibular third molars | day 7
  Early postoperative complications will be evaluated within the first postoperative week. Complications of interest include pain, facial swelling, trismus (limited mouth opening), prolonged bleeding, dry socket, infection at the surgical site, and neurosensory disturbances in the lower lip or chin region. At the postoperative day-7 visit, each complication will be recorded as present or absent based on clinical examination and patient report, and its severity will be classified descriptively (e.g. mild, moderate, severe). The proportion of patients experiencing each complication and any complication will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No